CLINICAL TRIAL: NCT05087160
Title: Socioeconomic Inequalities Exacerbates by Mitigation Measures Against COVID-19 in the Differential Prevalence of Prematurity and Low Weight in Uruguay
Brief Title: Socioeconomic Inequalities Exacerbated by Mitigation Measures to COVID-19 and Differences in Prematurity Prevalence
Status: Completed | Type: Observational
Sponsor: Universidad de la Republica (Other)
Responsible Party: Principal Investigator, Stephanie Viroga, Clinical professor, Universidad de la Republica
Other Study IDs: COVID-19 and perinatal results
Record Dates: First submitted 2021-10-06; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: COVID-19 Pandemic; Preterm; Low Birth-weight
Keywords: COVID-19; preterm; low birth weight
MeSH Terms: conditions — COVID-19; Premature Birth

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- semester pre pandemia in sub sectors of public health care in Uruguay: all birth in sub sectors of public health care between march 15 and September 30 of 2019, pre pandemia
- semester pre pandemia in sub sectors of private health care in Uruguay: all birth in sub sectors of private health care between march 15 and September 30 of 2019, pre pandemia
- semester with mitigation measures against COVID 19 in sub sectors of public health care in Uruguay: all birth in sub sectors of public health care between march 15 and September 30 of 2020, with mitigation measures against COVID- 19
  Interventions: Other: mitigation measures against COVID 19
- semester with mitigation measures against COVID 19 in sub sectors of private health care in Uruguay: all birth in sub sectors of private health care between march 15 and September 30 of 2020, with mitigation measures against COVID- 19
  Interventions: Other: mitigation measures against COVID 19

INTERVENTIONS:
Other: mitigation measures against COVID 19 — no intervention
  Groups: semester with mitigation measures against COVID 19 in sub sectors of private health care in Uruguay; semester with mitigation measures against COVID 19 in sub sectors of public health care in Uruguay

SUMMARY:
Objective: to assess the perinatal results in Uruguay during the semester of successful control of the COVID 19 pandemic to evaluate the impact of the crises in the public and private sub sectors of the Health System.

Methodology: An analytical observational study was carried out, comparing the semesters from March 15 to September 30, 2019 (year prior to the COVID 19 pandemic) with the same period 2020 (year of the COVID 19 pandemic), in the 2 sub sectors of public and private health care.

DETAILED DESCRIPTION:
An analytical observational study was carried out, comparing the semesters from March 15 to September 30, 2019 with the same period 2020, in the 2 sub sectors of public health care of the private sub sector throughout the country, taking all births in that period of time.

The semester selected is based on the fact that the first months of the pandemic were the ones with the greatest mitigation measures with drastic socio-economic consequences, but it was also a period of almost zero COVID infection in pregnancy, this being an opportune moment not to have as confounding factor to the maternal and fetal biological complications of this infection.

The situation will be analyzed in the 2 sub sectors of public health care, made up of the State Health Services Administration (ASSE), police health and military health, and the UDELAR Clinic Hospital, on the one hand, and the private sub-sector. made up of the Institutions of Collectivized Medical Assistance (IAMC) of Montevideo and the Interior (FEPREMI) and the private health care insurance.

The primary variable to be analyzed in both periods and in both subsectors of the national integrated system health was the incidence of preterm births (less than 37 weeks gestational age), low birth weight (newborns with a birth weight less than 2,500 grams) and intrauterine growth restriction (marked by doctor attending the birth, as a clinical diagnosis of the current pregnancy)

For the analysis of the national data, of the study periods, the database was requested from the Ministry of Public Health. This database is provided to researchers anonymously

ELIGIBILITY:
Inclusion Criteria:

* all live birth

Exclusion Criteria:

* stillbirth

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: all live births in the 2 sub sectors of public health care of the private sub sector in the selected period of time
Sampling Method: Non-Probability Sample
Enrollment: 37323 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
incidence of incidence of preterm births, low birth weight and intrauterine growth restriction | March 15 to September 30, 2019 and March 15 to September 30, 2020
  number of birth in total birth with these conditions en two periods time in the two subsectors of health care

CONTACTS AND LOCATIONS:
Locations (1):
- Stephanie Viroga, Montevideo, Uruguay

REFERENCES:
- [Derived] Briozzo L, Tomasso G, Trujillo J, Viroga S, Pintos J, Nozar F, Aleman A, Buekens P. COVID-19 mitigation measures increase preterm birth and low birth weight in the public healthcare system in Uruguay. Int J Gynaecol Obstet. 2023 Aug;162(2):718-724. doi: 10.1002/ijgo.14778. Epub 2023 Apr 13. PMID 37052316